CLINICAL TRIAL: NCT04460716
Title: Predictors for Postoperative Delirium After Major Noncardiac Surgery in Adults
Acronym: PODMAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Principal Investigator, Nicolai Goettel, Principal Investigator, University Hospital, Basel, Switzerland
Other Study IDs: PODMAS
Record Dates: First submitted 2020-06-25; First posted 2020-07-07 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Major noncardiac surgery — Vascular, thoracic, visceral, orthopedic, gynecologic, urologic, ENT, maxillo-facial, plastic and reconstructive surgery

SUMMARY:
This research project is an observational cohort study by retrospective chart review of patients that underwent major noncardiac surgery at University Hospital Basel, Switzerland, in the years 2011-2015. The PODMAS study aims to identify risk factors for POD in a general surgical population.

DETAILED DESCRIPTION:
The Diagnostic and Statistical Manual of Mental Disorders, 5th ed. (DSM-5) describes delirium as a "disturbance in attention (i.e., reduced ability to direct, focus, sustain, and shift attention) and awareness (reduced orientation to the environment)". In addition, a "disturbance in cognition (e.g., memory deficit, disorientation, language, visuospatial ability, or perception)" occurs. The deficits cannot be explained by other neurocognitive disorders.

Delirium develops within hours to a few days and can fluctuate in severity during the day. Acute delirium lasts a few hours or days, whereas persistent delirium lasts for weeks or months. In a hospital setting, delirium hardly ever lasts longer than a week but some symptoms can persist for months after the patient was discharged.

According to the International Statistical Classification of Diseases and Related Health Problems, 10th rev. (ICD-10), delirium is a pathologic brain disorder, which consists of a disturbance in consciousness, attention, perception, memory, psychomotor functions, emotional stability, and circadian rhythm. The severity can range from mild to very severe POD occurs in connection with a surgical procedure within the first four days after an intervention. 10-70% of all surgical patients above the age of 65 years are affected.

Delirium is not only a burden to the patient and their family by increasing functional and cognitive damages, and increasing mortality, it has a high impact on the economy, as well. A patient with delirium has a longer length of hospital stay, more complications, and often requires long-term care after being discharged from the hospital. All these aspects show the need for prevention of delirium.

There are various preoperative risk factors that influence the development of POD. Advanced age, preexisting cognitive impairment, depression and other psychopathologic symptoms, intake of psychotropic substances, sensory impairment like decrease in visual or auditory perception, impairment in daily life activities, dehydration, malnutrition, metabolic dysfunctions, urinary catheters, severe diseases and different comorbidities such as chronic cardiac insufficiency, atrial fibrillation, or previous history of stroke or infections favor the development of delirium.

The incidence of POD after major noncardiac surgery and the burden to patients and healthcare systems in general is high.

This research project is an observational cohort study by retrospective chart review of patients that underwent major noncardiac surgery at University Hospital Basel, Switzerland, in the years 2011-2015. The PODMAS study aims to identify risk factors for POD in a general surgical population.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent major noncardiac surgery at the University Hospital Basel during the years 2011-2015.

Exclusion Criteria:

* Patients that died during the operation or one day after surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent major noncardiac surgery at the University Hospital Basel during the years 2011-2015.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Daily assessment of postoperative delirium from postoperative day 1 up to postoperative day 30 or hospital discharge, whichever comes first
  Incidence of postoperative delirium assessed by a validated delirium measurement tool (CAM, 3D-CAM, CAM-ICU, ICDSC, MDAS, GAR, DOSS, Nu-DESC, DRS-R-98, and/or patient chart review)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolai Goettel, MD, Principal Investigator — University Hospital, Basel, Switzerland